CLINICAL TRIAL: NCT03947008
Title: The Effects of Intuitive Eating on Body Appreciation and Dietary Restraint in College Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carly R Pacanowski (Other)
Collaborators: University of Delaware (Other)
Responsible Party: Sponsor-Investigator, Carly R Pacanowski, Faculty Support, University of Delaware
Organization: University of Delaware (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1346035-1
Record Dates: First submitted 2019-01-09; First posted 2019-05-13 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Eating Behavior; Body Image; Dietary Habits; Restricted Behavior
Keywords: intuitive eating; dietary restraint
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: The proposed pilot study will evaluate the feasibility and acceptability of an intuitive eating program for University of Delaware college women. A randomized controlled design will be used to study the effects of an intuitive eating intervention on body dissatisfaction and dietary restraint in young adult women, thereby reducing risk of eating disorders. There will be 2 arms of this study. The First Intuitive Eating Group (IE1) will act as the intervention group and receive the intervention first. The Second Intuitive Eating Group (IE2) will act as a waitlist group and receive the intervention the week immediately following the end of IE1's course.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Intuitive Eating Group (IE1) (Experimental): IE1 will be the first group to participate in an intuitive eating program and will be required to attend five intuitive eating classes. The intuitive eating classes will be 60-minutes each week for 5 weeks. An initial assessment will be conducted during the first thirty minutes of the first intuitive eating class. A final assessment will be conducted during the last 30 minutes of the last intuitive eating class. This group will have an additional final assessment on the last day of the IE2's intuitive eating course. During the assessments, they will complete a questionnaire that will ask them about their body satisfaction and eating attitudes, and have their height and weight measured.
  Interventions: Other: Intuitive Eating Program
- Second Intuitive Eating Group (IE2) (Experimental): IE2 will be the second group to will participate in an intuitive eating program and will be required to attend 5 intuitive eating classes. The classes will be 60-minutes each week for 5 weeks. An initial assessment will be conducted on the same day as IE1 but they will take the 5 week course once the first group completes the class. This group will have an additional initial assessment on the day they begin their curriculum. The initial assessment will occur during the first thirty minutes of the first intuitive eating class. A final assessment will be conducted during the last 30 minutes of the last intuitive eating class. During assessments, they will complete a questionnaire that will ask about body satisfaction and eating attitudes, and have their height and weight measured.
  Interventions: Other: Intuitive Eating Program

INTERVENTIONS:
Other: Intuitive Eating Program — A 5-week Intuitive Eating Curriculum created by a Registered Dietitian, Kaylee Frazier, will be used. The creator of this curriculum was contacted for permission and the curriculum was modified for use with college women.
  The goal of the program is to challenge and eventually shift participant's mindset from the traditional diet culture towards a way of eating that is driven by their unique bodily needs. Content will focus on training participant to listen to their internal body cues for hunger opposed to restricting or eliminating foods. A list of intuitive eating principles and ways to incorporate them into daily routines will be provided to the participants throughout the sessions, coupled with homework assignments, journaling, and exercises to be completed before subsequent sessions.

SUMMARY:
College-aged women are at risk for eating disorders and disordered eating, which present serious health concerns. Two potent risk factors for eating disorders, body dissatisfaction and dietary restraint, are common among female college students.

Intuitive eating is a strategy in which instead of listening to the predominant 'diet culture' and focusing on things like calories and energy balance, individuals practice listening to their internal physiological signals to decide when and what to eat and when to stop. Based on current research, intuitive eating has been shown to foster body satisfaction and healthy eating attitudes among women.

The proposed pilot study will evaluate the feasibility and acceptability of an intuitive eating program for University of Delaware college women. In addition, this study will test the hypothesis that the intuitive eating program will reduce cognitive factors of body dissatisfaction and dietary restraint in females compared to a waitlisted group. Additionally, the investigators expect this reduction in dietary restraint to be associated with less disordered eating behavior. Exploratory aims include measuring engagement in disordered eating behaviors and changes in weight over the study period. This preliminary data will be used to estimate effect sizes for larger future trials.

DETAILED DESCRIPTION:
The overall goal of the program is to challenge and eventually shift participant's mindset from the traditional diet culture towards a way of eating that is driven by their unique bodily needs. Thus, content will focus on training participant to listen to their internal body cues for hunger opposed to restricting or eliminating foods. A list of intuitive eating principles and ways to incorporate them into daily routines will be provided to the participants throughout the sessions, coupled with homework assignments, journaling, and exercises to be completed before subsequent sessions.

This program will be delivered by two Registered Dietitians from the University of Delaware, Julia Katcher and Maryann Eastep. Both will have received training from https://www.helmpublishing.com/intuitive-eating-certificate-of-training-1891 and will have become Certified Intuitive Eating Counselors by the start of Spring 2019.

After being screened for eligibility and meeting eligibility criteria, the individual will be emailed by the PI, who will invite the individual to participate in the study and enclose an invitation for their first intuitive eating class. This email will also include a copy of the consent form for them to review and decide if they want to commit to the study. If the individual is still interested in participating they will email the PI again to be placed on the participant list. After 24 individuals, who have met screening criteria, have indicated desire to participate, they will be randomized to one of two conditions: (1) First Intuitive Eating Group (IE1) offered once per week for 5 weeks; or (2) Second Intuitive Eating Group (IE2), who will receive the same intuitive eating course after the first group has concluded.

Baseline assessments will be conducted on all participants, both IE1 and IE2, on the same day, at the beginning of the first intuitive eating class for IE1 group. These assessments will be conducted by the project staff identified above. The assessment should not take longer than 30 minutes. When the participants arrive, they will first have the opportunity to discuss the study with the PI, ask any questions or address any concerns they might have and if interested, sign the consent form. Consent forms will be provided, prior to the initial assessment and the intuitive eating class beginning, to be reviewed and signed in the presence of the PI.

After signing the consent form, then they will fill out the questionnaire. The investigators will measure attitudes about body satisfaction and eating.

Lastly, the individuals will have their questionnaires checked by a member of the research team to ensure completion. After signing the consent form and turning in their questionnaires, participants will receive their group assignment. They will either be assigned to the first intuitive eating group (IE1) or the second intuitive eating group (IE2).

If they were assigned to the IE1 group, they will complete their first class immediately following the baseline assessment at the beginning of the Spring 2019 semester.

If they are assigned to the IE2 group, they will complete their first intuitive eating class the week after IE1's 5-week intuitive eating course has been completed.

Each group will be able to attend up to 5 intuitive eating sessions that are 60 minutes long for a total of 5 weeks. Participation in the intuitive eating program will be tracked by documenting presence or absence at each intuitive eating session. A member of the research team will be responsible for documenting this and also checking fidelity to the curriculum.

An additional baseline assessment will be conducted on the IE2 Group at the beginning of their first intuitive eating class. This assessment protocol will be identical to the one they attended, as described above, on the first day the IE1 group began their intuitive eating course. The assessment should not take longer than 30 minutes.

End-of-study assessments will be completed on the last day of the participant's intuitive eating program. The assessment should not take longer than 30 minutes. At the last intuitive eating classes for each session, the investigators will measure attitudes about body satisfaction and eating, height, and weight.

A program evaluation survey will be passed out during the end of the last intuitive eating class for both IE1 and IE2. This is to assess the effectiveness of the intuitive eating program and to receive feedback from participants on where the investigators can improve this program. This program evaluation is included with this application.

IE1 will be asked to come back for an additional final assessment and feedback session on the last session day of IE2's intuitive eating course. IE1 will be in a separate room where they will have the chance to discuss and provide program feedback to the Graduate and Undergraduate Research Assistants. They will also fill out a program evaluation survey (for the second time), as described above. IE2 will be in the room where their last session just concluded where they will fill out the final survey, as described above, and will have their height and weight measured. Once both groups are finished in each room, they will switch and go through the same protocol as the last group did in that room

ELIGIBILITY:
Inclusion Criteria:

* The participant is between the age of 18-26;
* University of Delaware student;
* Willing and able to commit to the 5-week study at specified time;
* Has a history of body dissatisfaction as indicated by high survey scores on body satisfaction and high scores on dietary restraint; and
* Are not currently being treated for an eating disorder.

Exclusion Criteria:

* Females who are currently diagnosed with and/or seeking treatment for an eating disorder.

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Dietary Restraint | 5 weeks
  Measured via a survey that uses questions from the following validated questionnaires:
  ●Three-Factor Eating Questionnaire-18
  * Measures dietary restraint
  * Means are computed for three subscales and are transformed to a 0-100 scale score
  * Higher scores indicate greater cognitive restraint, uncontrolled, emotional eating
Body Appreciation: survey | 5 weeks
  Body appreciation will be measured via a survey. This survey uses questions from the validated Body Appreciation Scale-2. There are 10 questions rated from 1 "never to 5 "always". The 10 scores from each question are totaled and averaged. Higher scores reflect greater body appreciation.
Intuitive Eating | 5 weeks
  Measured using the following validated survey:
  ●Intuitive Eating Scale - 2
  * Measures tendency to follow physical hunger and fullness cues
  * *Total*score range = 5-115
  * Higher scores indicate greater levels of intuitive eating or its dimensions
Interoceptive Awareness | 5 weeks
  Measured using the Multi-Dimensional Assessment of Interoceptive Awareness -2

SECONDARY OUTCOMES:
Weight | 5 weeks
  Weight will be measured using a research-grade body weight scale. There will be a measurement station run by trained anthropometrists. The station will be enclosed by a divider to ensure privacy. Weight will be taken in light clothing, with shoes removed, twice, and rounded to the nearest tenth of a kg.
Height | 5 weeks
  Height will be measured using a stadiometer. There will be a measurement station run by trained anthropometrists. The station will be enclosed by a divider to ensure privacy. Height will be taken twice, rounded to the nearest cm.

CONTACTS AND LOCATIONS:
Overall Officials: Carly Pacanowski, PhD, Study Director — Faculty Support
Locations (1):
- University of Delaware, Newark, Delaware, United States